CLINICAL TRIAL: NCT04037462
Title: Induction of Sensecence Using Dexamethasone to Re-sensitize NSCLC to Anti-PD1 Therapy
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Wayne State University (Other); University of Michigan (Other); Barbara Ann Karmanos Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSDR-002-18F
Record Dates: First submitted 2019-07-26; First posted 2019-07-30 (Actual); Results first posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-05

CONDITIONS: Non-Small Cell Lung Cancer; Immunotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: In the first stage, three Dex escalation cohorts will be evaluated sequentially from Cohort A to Cohort C until > 2 patients exhibit FLT-PET response (i.e., 30% reduction in FLT-PET uptake in at least one target lesion); otherwise, the trial will be terminated due to futility. The secondary objective is to assess the effect of Dex on pembrolizumab in terms of overall response rate (ORR).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lead in Dexamethasone followed by immunotherapy (Experimental): escalating doses of pretreatment dexamethasone in patients who have failed initial immunotherapy to 1. assess changes in FLT PET uptake 2. assess overall response rates of pretreatment dexamethasone (dose from 1) on subsequent immunotherapy re-challenge
  Interventions: Drug: Dexamthasone

INTERVENTIONS:
Drug: Dexamthasone — escalating doses of pretreatment dexamethasone in patients who have failed initial immunotherapy to 1. assess changes in FLT PET uptake 2. assess overall response rates of pretreatment dexamethasone (dose from 1) on subsequent immunotherapy re-challenge

SUMMARY:
Lung cancer accounts for 30% of all cancers among American war Veterans and remains the leading cause of cancer related deaths. Half of all lung cancers are metastatic non-small cell lung cancer (NSCLC), with a 2-year survival rate of 10%. Immunotherapy with immune checkpoint inhibitors (ICI) has emerged as a promising therapeutic strategy that aims to harness the immune system to fight lung cancer. However, given the modest response rates of 20-25% to these immune checkpoint inhibitors, there is a greater desire to extend their benefits to more patients. Along with the desire to extend their benefits, there is a critical need for the development of novel approaches that can expand the benefit from immune checkpoint inhibitors and create more durable responses, prolonging survival from lung cancer. The investigators' studies show that extended dexamethasone (Dex) treatment induces irreversible cell cycle blockade and a senescence phenotype through chronic activation of the p27Kip1 gene in glucocorticoid receptor (GR) overexpressing lung adenocarcinoma (AC) cell populations. Further, following withdrawal of Dexamethasone, proteins associated with the senescence associated secretory phenotype (SASP) strongly attracted and expanded T-cells, NK cells and monocytes stimulated tumor cell cytolytic activity of NK cells. Therefore, dexamethasone may induce a persistent senescence phenotype in tumor cell sub-populations expressing moderate/high levels of GR and resultant chemokines produced by the senescent cells will mobilize host immune cells to reboot response to immune checkpoint inhibitors following complete Dexamethasone withdrawal.

DETAILED DESCRIPTION:
Lung cancer accounts for 30% of all cancers among American war Veterans and remains the leading cause of cancer related deaths. Half of all lung cancers are metastatic non-small cell lung cancer (NSCLC), with a 2-year survival rate of 10%. Immunotherapy with immune checkpoint inhibitors (ICI) has emerged as a promising therapeutic strategy that aims to harness the immune system to fight lung cancer. However, given the modest response rates of 20-25% to these immune checkpoint inhibitors, there is a greater desire to extend their benefits to more patients. Along with the desire to extend their benefits, there is a critical need for the development of novel approaches that can expand the benefit from immune checkpoint inhibitors and create more durable responses, prolonging survival from lung cancer.

Our studies show that extended dexamethasone (Dex) treatment induces irreversible cell cycle blockade and a senescence phenotype through chronic activation of the p27Kip1 gene in glucocorticoid receptor (GR) overexpressing lung adenocarcinoma (AC) cell populations. Further, following withdrawal of Dexamethasone, proteins associated with the senescence associated secretory phenotype (SASP), particularly CCL2, CCL4, CXCL1 and CXCL2 strongly attracted and expanded T-cells, NK cells and monocytes stimulated tumor cell cytolytic activity of NK cells.

Our overarching hypothesis is that in lung adenocarcinoma patients who are not on baseline steroids, pre-treatment with Dexamethasone will induce a persistent senescence phenotype in tumor cell sub-populations expressing moderate/high levels of GR and resultant chemokines produced by the senescent cells will mobilize host immune cells to reboot response to immune checkpoint inhibitors following complete Dexamethasone withdrawal. The investigators will test this hypothesis through the conduct of the following aims.

Specific Aim 1: Use FLT-PET imaging and blood analysis to test whether a 7-14-day pre-treatment of lung adenocarcinoma patients with Dexamethasone followed by Dexamethasone withdrawal will induce persistent senescence related cell cycle arrest in 1 lesion in 60% of patients, (based on GR expression) accompanied by release of SASP proteins and activation of T and NK cells.

Specific Aim 2: Test whether a 7-14-day pre-treatment of lung adenocarcinoma patients with Dexamethasone followed by Dexamethasone withdrawal and subsequent re-challenge with pembrolizumab will yield an overall response rate (ORR) of 33% to pembrolizumab in association with tumor GR status, SASP and immune cell activation.

These aims will be conducted through a Phase II clinical trial designed as a single-arm two-stage study in Veterans whose lung adenocarcinoma has progressed on immune checkpoint inhibitors. Based on the investigators' preliminary data, the investigators expect that Dexamethasone will induce tumor senescence in at least one lesion in 60% of patients and secondarily improve overall response to pembrolizumab by 33%. Success with these aims would inform a larger study that could potentially change the way the investigators approach patients with primary or acquired resistance to immune checkpoint inhibitors with an off the shelf medication that could re-sensitize lung adenocarcinoma to immune checkpoint inhibitors. The proposed research could substantially benefit Veterans with metastatic NSCLC, a group with the most genomically complex lung cancers and poor survival.

ELIGIBILITY:
Inclusion Criteria:

* Be willing and able to provide written informed consent/assent for the trial.
* Be 18 years of age on day of signing informed consent.
* Have a life expectancy of at least 6 months.
* Have a histologically confirmed diagnosis of stage IV NSCLC (includes patients who have progressed on durvalumab for Stage III NSCLC) and have at least one measurable lesion based on RECIST v1.1.
* Have a performance status of 0, 1 or 2 on the ECOG Performance Scale (Appendix 15.1).
* Demonstrate adequate organ function all screening labs should be performed within 14 days of enrollment.
* Female subject of childbearing potential should have a serum pregnancy within 14 days of enrollment and 72 hours prior to receiving the first dose of study medications.
* Female subjects of childbearing potential must be willing to use a highly effective method of contraception as outlined in Section 6.3.3 for the course of the study through 180 days after the last dose of study medications.

  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Male subjects of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 180 days after the last dose of study therapy.

  * Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Adequate tissue sample for correlative studies. A new sample is not necessary if archival specimen is available and has adequate amount of tumor content (at least 30%). This needs to be determined by a pathologist.

Exclusion Criteria:

* Received palliative radiation within 7 days of enrollment.
* Has a known history of prior malignancy except if the patient has undergone potentially curative therapy with no evidence of that disease recurrence for 5 years since initiation of that therapy.

  * Note: the time requirement for no evidence of disease for 5 years does not apply to the NSCLC tumor for which a subject is enrolled in the study. The time requirement also does not apply to subjects who underwent successful definitive resection of basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to enrollment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior enrollment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Has active autoimmune disease that has required systemic treatment within the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs).

  * Note: Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Subjects requiring daily corticosteroids >10mg of prednisone (or its equivalent) would be excluded from the study.

  * Note: Subjects with asthma that require intermittent use of bronchodilators, inhaled steroids, or local steroid injections would NOT be excluded from the study.
* Has evidence of interstitial lung disease or a history of non-infectious pneumonitis that required oral or intravenous glucocorticoids to assist with management.

  * Note: Lymphangitic spread of the NSCLC is not exclusionary.
* Has an active infection requiring systemic therapy.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* Subjects with cognitive functioning/impairment based on medical record review ad physician decision.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with informed consent through 180 days after the last dose of trial treatment.
* Has a diagnosis of immunodeficiency (including Human Immunodeficiency Virus (HIV) or acquired immunodeficiency (AIDS)-related illness) or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to enrollment.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has known active Hepatitis B or Hepatitis C.
* Has received a live vaccine within 30 days of enrollment.

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.
* BASELINE CORTICOSTEROID AT STUDY ENTRY - subjects may not be on any steroids (dexamethasone, prednisone, etc) at the time of consent/study start.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-07-07 (Actual); Primary Completion 2022-02-23 (Actual); Study Completion 2023-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nithya Ramnath, MD, Principal Investigator — VA Ann Arbor Healthcare System, Ann Arbor, MI
Locations (1):
- VA Ann Arbor Healthcare System, Ann Arbor, MI, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment start date July 7, 2021, consented 3 participant from the medical oncology clinic. 1 participant rescinded consent and was never enrolled therefore, we only enrolled 2 participants start shut down during COVID 2020-21 Pt 1: 7-7-2021 Pt 2: 8-30-2021 (rescinded consent due to logistical burden) Pt 3: 1-05-2022
Pre-assignment Details: Pt 2 rescinded consent due to logistical burden
Groups:
- Lead in Dexamethasone Followed by Immunotherapy: lead in cohort consisted of patients who failed initial immunotherapy and were assigned to dose level 1: dexamethasone 4 mg p.o b.i.d days 1-7 to assess 1. changes in FLT PET uptake 2. assess overall response rates of pretreatment dexamethasone on subsequent immunotherapy re-challenge.
Period: Overall Study
Arm/Group | Lead in Dexamethasone Followed by Immunotherapy
Started | 2 (Study closed on 11-29-22 due to poor accrual after 1 evaluable pt was accrued. Therefore, initial milestones were not achieved)
Completed | 2 (Only 1 pt (Pt 1) was evaluable. On 1st response evaluation on 9-15-21 had progressive disease and came off study)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Lead in Dexamethasone Followed by Immunotherapy
Number analyzed (Participants) | 2
Age, Customized [Number; unit: years]
  greater than or equal to 18 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in Fluoro-3' Deoxythymidine Positron Emission Tomography (FLT-PET) Signal
Description: In the first stage, three Dex escalation cohorts will be evaluated sequentially from Cohort A to Cohort C until > 2 patients exhibit FLT-PET response (i.e., 30% reduction in FLT-PET uptake in at least one target lesion); otherwise, the trial will be terminated due to futility.
  The SUVmax will be measured at baseline and after Dex run-in and wash out period. For example, in Cohort A, patients will get an FLT- PET at baseline, then receive Dexamethasone 4mg PO BID given for 7 days, followed by taper over 2-4 days and 3 day wash out and then the post-Dex FLT-PET.
Time Frame: Baseline and Post DEX (14 days)
Measure: Mean (Standard Deviation); unit: SUVmax
Groups:
- Lead in Dexamethasone Followed by Immunotherapy: escalating doses of pretreatment dexamethasone in patients who have failed initial immunotherapy to 1. assess changes in FLT PET uptake 2. assess overall response rates of pretreatment dexamethasone (dose from 1) on subsequent immunotherapy re-challenge
  Dexamthasone: escalating doses of pretreatment dexamethasone in patients who have failed initial immunotherapy to 1. assess changes in FLT PET uptake 2. assess overall response rates of pretreatment dexamethasone (dose from 1) on subsequent immunotherapy re-challenge
  Due to accrual of 2 participants there is not enough data to state efficacy.
Arm/Group | Lead in Dexamethasone Followed by Immunotherapy
Number analyzed (Participants) | 2
SUVmax
  Baseline | 6.63 (.95)
  Post DEX | 6.05 (1.24)

2. Secondary Outcome: Response Rate
Description: The primary objective in SA 2 is to assess the effect of Dex on pembrolizumab in terms of overall response rate (ORR). Based on pre-clinical and clinical studies, the investigators hypothesize that the true ORR of Dex followed by pembrolizumab will be at least 33% (i.e., p1 = 0.33) vs. the historical control whose ORR is at most 7% (i.e., p0 = 0.07). The ORR will be statistically evaluated when the FLT-PET response trial enters the third stage, where the number of patients with the selected optimal Dex duration will be 21. Otherwise, ORR will be summarized descriptively. The null hypothesis (p0 = 7%) will be rejected if five or more responses are observed in 21 patients, which yields a 1-sided type I error rate of 5% and power of 87% when the true ORR is 33% (i.e. p1 = 33%).
Time Frame: 3 months
Population: Overall response rate will be assessed at 12 week FDG PET scan
Measure: Count of Participants; unit: Participants
Arm/Group | Lead in Dexamethasone Followed by Immunotherapy
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Time Frame: 1 Year
Arm/Group | Lead in Dexamethasone Followed by Immunotherapy
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
We consented 3 participants and had one subject rescind consent leaving us with 2 enrolled participants. of the 2 participants only was was evaluable. Therefore, we do not have sufficient data to prove outcomes measures

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-07-21): https://cdn.clinicaltrials.gov/large-docs/62/NCT04037462/Prot_SAP_001.pdf
  • Informed Consent Form (2020-11-12): https://cdn.clinicaltrials.gov/large-docs/62/NCT04037462/ICF_000.pdf